CLINICAL TRIAL: NCT01807377
Title: A Phase 1 Placebo-Controlled Study To Assess Safety, Tolerability, Pharmacokinetics And Effect On Midazolam Pharmacokinetics Of Multiple Oral Doses Of PF-05175157 Administered In A Tablet Formulation In Otherwise Healthy Overweight And Obese Subjects
Brief Title: Multiple Dose Safety Tolerability, Pharmacokinetics And Midazolam Interaction In Healthy Overweight And Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B1731021
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-05175157, Midazolam (Experimental): Day 0: Midazolam 2 mg administered alone Days 1-14: 200 mg PF-05175157 administered BID Day 11: Midazolam and PF-05175157
  Interventions: Drug: PF-05175157; Drug: Midazolam
- Placebo, Midazolam (Experimental): Day 0: Midazolam 2 mg administered alone Days 1-14: Placebo administered BID Day 11: Midazolam and Placebo
  Interventions: Other: Placebo; Drug: Midazolam

INTERVENTIONS:
Drug: PF-05175157 — 200 mg tablet administered twice per day for 14 days
  Arms: PF-05175157, Midazolam
Drug: Midazolam — 2mg administered as single doses on Days 0 and 11
  Arms: PF-05175157, Midazolam
Other: Placebo — Placebo administered twice per day for 14 days
  Arms: Placebo, Midazolam
Drug: Midazolam — 2mg administered as single doses on Days 0 and 11
  Arms: Placebo, Midazolam

SUMMARY:
This study is designed to assess the safety, tolerability and pharmacokinetics of multiple oral 200-mg doses of PF-05175157 administered twice daily for 14 days in healthy overweight and obese subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Women must be of non childbearing potential.
* Body Mass Index (BMI) of 25 to 35 kg/m2 inclusive; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Evidence or history of any chronic ongoing or current pulmonary disease.
* History of smoking in the past 5 years and a history of smoking more than 10 pack years, or history or evidence of habitual use of other (non smoked) tobacco or nicotine containing products. Active ocular disease including infection, glaucoma, seasonal allergies, dry eye symptoms or retinal/optic nerve disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma PF-05175157 Concentration (Cmax) | 0 - 10 hrs postdose
  Single Dose
Area Under the Curve from Time Zero to end of dosing interval for PF-05175157 (AUCtau) | 0 - 10 hrs postdose
  Single Dose
Time to Reach Maximum Observed Plasma PF-05175157 Concentration (Tmax) | 0 - 10 hrs postdose
  Single Dose
Maximum Observed Plasma PF-05175157 Concentration (Cmax) | 0 - 48 hours postdose
  Steady State
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) for PF-05175157 | 0 - 48 hours postdose
  Steady State
Time to Reach Maximum Observed Plasma PF-05175157 Concentration (Tmax) | 0 - 48 hours postdose
  Steady State
Apparent Oral Clearance of PF-05175157 (CL/F) | 0 - 48 hours postdose
Accumulation Ratio of PF-05175157 (Rac) | 0 - 10 hours postdose
Plasma Decay Half-Life of PF-05175157 (t1/2) | 0 - 48 hours postdose
Apparent Volume of Distribution of PF-05175157 (Vz/F) | 0 - 48 hours postdose
Urinary Recovery for PF-05175157 (AE24) | 0 - 24 hours postdose
  Amount of PF-05175157 recovered in urine over 24 hours
Renal Clearance for PF-05175157 (CLr) | 0 - 24 hours post dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration for midazolam [AUC (0-t)] | 0 - 48 hours postdose
Area Under the Curve From Time Zero to Extrapolated Infinite Time for midazolam [AUC (0 - inf)] | 0 - 48 hours postdose
Maximum Observed Plasma Concentration for midazolam (Cmax) | 0 - 48 hours postdose
Time to Reach Maximum Observed Plasma midazolam Concentration (Tmax) | 0 - 48 hours post dose
Plasma Decay Half-Life of midazolam (t1/2) | 0 - 48 hours postdose
Fasting triglycerides | 14 days
Total cholesterol | 14 days
LDL cholesterol | 14 days
HDL cholesterol | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Chula Vista, California, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1731021&StudyName=Multiple%20Dose%20Safety%20Tolerability%2C%20Pharmacokinetics%20And%20Midazolam%20Interaction%20In%20Healthy%20Overweight%20And%20Obese%20Subjects%0A